CLINICAL TRIAL: NCT03747887
Title: Enhancing IEPs of Children With ADHD Using Daily Report Cards: An Efficacy Trial
Brief Title: Enhancing IEPs of Children With ADHD Using Daily Report Cards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Florida International University (Other)
Responsible Party: Principal Investigator, Gregory Fabiano, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A180175
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Schools

STUDY DESIGN:
Intervention Model Description: Random assignment to intervention group or business as usual group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School as Usual (Active Comparator): School as usual comparison condition.
  Interventions: Other: School as Usual
- Daily Report Card (Experimental): A coach will establish a Daily Report Card based on IEP goals and objectives with the parents/teachers of the child in this arm.
  Interventions: Behavioral: Daily Report Card

INTERVENTIONS:
Behavioral: Daily Report Card — Students assigned to the DRC group will have a consultant assigned to the student for the duration of the school year. The consultant will work with the child's primary special education teacher (or regular education teacher if the child spends the majority of his or her day mainstreamed) to establish a DRC over the course of three consultation visits. The How to Establish a Daily Report Card manual contains a standard DRC instruction packet that is provided to teachers to explain the rationale of the DRC, procedures for creating, modifying, and evaluating the DRC, procedures for parents to create home-based rewards for DRC performance, and information on trouble-shooting.
  Arms: Daily Report Card
Other: School as Usual — The Individualized Education Program will be implemented as usual, with no additional study-related supports.
  Arms: School as Usual

SUMMARY:
The purpose of this study are to determine the effectiveness of the daily report card (DRC) approach to supporting children with ADHD in special education in schools compared to a business as usual condition. Children in the study will be randomly assigned to business as usual, or to receive a DRC based on Individualized Education Program goals and objectives, across the school year. All children will have progress carefully monitored across the school year.

DETAILED DESCRIPTION:
This study will investigate the efficacy of an intervention to enhance the special education supports used for children with ADHD (i.e., the manner in which goals/objectives on the IEP are monitored and addressed; targeting of social/behavioral goals).

The purpose of this proposed study is to provide evidence for the efficacy of using a daily report card intervention (DRC) as a means of linking the child with ADHD's IEP goals and objectives to his/her daily functioning in the classroom environment. A Goal 2 study was recently completed to develop and provide preliminary support for the DRC intervention for this purpose (Fabiano et al., 2010). The proposed investigation will be a multi-site study conducted in elementary schools throughout the Western New York and South Florida area. Participants will be 216 children (grades K-6), who have been diagnosed with ADHD and have an IEP (e.g., Specific Learning Disability, Emotionally Disturbed, Other Health Impaired).

In the proposed study, the efficacy of the DRC as an enhancement to children with ADHD's IEPs will be investigated in an experimental study. Children will be randomly assigned on the individual level to a condition where a behavioral consultant works with the child's teacher(s) to construct a DRC, implement it, and monitor it, or to an IEP only, school as usual (SAU) condition, where teachers will attempt to meet the IEP goals and objectives as they typically would. A DRC is an operationalized list of target behaviors (e.g., "completes reading assignments with 80% accuracy or better," "has no office time outs during the day") that are evaluated each day by the teacher. The DRC is used as a means of providing the child and parent feedback on progress on a daily basis, and it doubles as a mechanism teachers can use to track and monitor the child's behavior and progress on key functional domains. The DRC can be easily linked to IEP goals and objectives, providing a bridge between the IEP and the child's daily functioning in the classroom. Parents will also be taught in parenting meetings how to reward their child at home for successful attainment of DRC goals and how to communicate effectively with their child's teacher.

Measures of key outcomes will include observations of behavior in the classroom conducted by observers naïve to group assignment or study hypotheses, academic performance outcomes, parent and teacher ratings of functioning, and IEP goal attainment. Primary measures of outcome will be analyzed using ANCOVA procedures. Secondary measures will include teacher ratings of ADHD and disruptive behavior/impairment. Additional analyses will investigate moderators (grade level, comorbid aggressive behavior, IEP quality). It is further hypothesized that classroom environment and fidelity of implementation at school/home will mediate outcomes (i.e., classroom climate, the fidelity of teacher monitoring/feedback regarding behavior, consistency of parent-implemented consequences at home).

ELIGIBILITY:
Inclusion Criteria:

* Current Individualized Education program
* Diagnosis of ADHD
* Enrolled in Grades Kindergarten - 6

Exclusion Criteria:

* IQ < 70
* Home-schooled
* Enrolled in a classroom with another study participant
* Autism spectrum disorder

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Student Behavior Teacher Response Observation Rule Violations Count | 5 months
  Frequency count of classroom rule violations collected during three, 30-minute observation periods and averaged.

SECONDARY OUTCOMES:
Academic Performance Rating Scale | 5 months
  Academic Performance Rating Scale sub scales of: Academic Productivity factor (7 items) that relates to work completion and accuracy, independent work, and following directions (coefficient alpha = .94; test-retest reliability over two weeks = .93), and an Academic Success (12 items) factor related to the child's academic achievement, recall, and ability (coefficient alpha = .95; test-retest reliability over two weeks = .91). Items are rated by teachers on a five-point Likert scale, and scores are summed for each of the two factors. Scores range from 5-35 for the Academic Success factor and from 5-60 for the Academic Productivity factor. Higher scores are representative of stronger classroom functioning
IEP Goals/Objectives met | 5 months
  Teacher rating at endpoint of goals/objectives met on an improvement rating scale ranging from very much worse to very much better. Scores across goals/objectives will be averaged for a single overall score, and higher scores indicated greater degrees of goal attainment.
Impairment rating scale - teacher version | 5 months
  Ratings of functional impairment on a 7-point visual analogue scale ranging from 0-6. Lower ratings indicated less impairment in functioning in each domain. Scores across domains will be averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
At the completion of the study, an anonymous database will be created and shared as per the data sharing plan constructed as part of the grant.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the completion of the study in 2021.
Access Criteria: Contact Dr. Fabiano directly at fabiano@buffalo.edu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03747887/Prot_SAP_000.pdf